CLINICAL TRIAL: NCT04711850
Title: A Prospective, Observational Long-term Follow-up Trial of Kidney Transplant Patients Treated With Imlifidase or Plasma Exchange After an Active/Chronic Active Antibody-Mediated Rejection Episode
Brief Title: An Long-term Follow-up Trial of Kidney Tx Patients Treated With Imlifidase or PE After an AMR
Status: Terminated | Type: Observational
Why Stopped: This is an internal decision based on prioritisations and no safety issues have been raised during the trial.
Sponsor: Hansa Biopharma AB (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-HMedIdes-18; 2020-004777-49 (EudraCT Number)
Record Dates: First submitted 2021-01-13; First posted 2021-01-15 (Actual); Results first posted 2025-05-11 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Kidney Transplant Rejection
MeSH Terms: interventions — Mac-1-like protein, Streptococcus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples collected for DSA and ADA may be stored for a maximum of 5 years after completion of the trial.
  A full chain of custody is maintained for all samples throughout their life cycle.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Imlifidase treatment in feeder Study 16-HMedIdeS-12: No treatment is given in this long-term follow-up study. In the feeder study (16-HMedIdeS-12) the patients in this group were treated with imlifidase.
  Interventions: Drug: Imlifidase
- Plasma exchange (PE) treatment in feeder Study 16-HMedIdeS-12: No treatment is given in this long-term follow-up study. In the feeder study (16-HMedIdeS-12) the patients in this group were treated with PE.

INTERVENTIONS:
Drug: Imlifidase — Immunoglobulin G degrading enzyme of Streptococcus pyogenes
  Other Names: IdeS, HMED-IdeS
  Groups: Imlifidase treatment in feeder Study 16-HMedIdeS-12

SUMMARY:
The aim of this trial is to collect data and provide a better understanding of the long-term outcome of imlifidase treatment on active or chronic active antibody-mediated rejection (AMR) in kidney transplant recipients. This is done by collecting data during an extended follow-up period of 3 years of clinical study trial 16-HMedIdeS-12, in which patients received either imlifidase or plasma exchange (PE) as AMR treatment. Data for parameters such as kidney graft survival, patient survival, kidney function, treatment of rebound of donor specific antibodies (DSA) and anti-drug antibodies (ADAs) are collected.

DETAILED DESCRIPTION:
AMR is one of the most challenging adverse events following kidney transplantation and a major cause of graft dysfunction and graft loss. AMR is triggered by donor-specific antibodies (DSA).Transplant glomerulopathy is a known consequence of persistent DSA positivity which results in graft failure and return to dialysis with attendant consequences for the patient and financial costs for the health care system.

The time from transplantation to onset of clinical symptoms of AMR varies largely between individuals. An early AMR (<30 days post-transplant) is commonly classified as active AMR and most often triggered by an immunological recall response with pre-existing DSA. A late AMR (>30 days post-transplant) is classified as either active or chronic active AMR and is caused by either a recall DSA response or newly developing naïve immune response associated with de novo DSA production.

There is no currently approved therapy for AMR and patients are often treated with a combination of therapies i.e., high dose IVIg +/- rituximab, PE with low dose IVIg +/- rituximab, and eculizumab which makes analysis of efficacy of any single agent difficult. Hence, there is a large unmet clinical need for new therapies to treat AMR.

Imlifidase is an IgG-degrading enzyme of Streptococcus pyogenes that cleaves all four human subclasses of IgG with high efficacy and specificity. The rapidity of the IgG cleavage by imlifidase is considered a major advantage as compared with PE, which often requires several rounds over several days to achieve a sufficient DSA reduction. Within a few hours after imlifidase dosing, the entire pool of IgG is completely cleaved and thereby a window where IgG levels are kept very low for approximately one week is created.

The short-term efficacy and safety of imlifidase in active and chronic active AMR is being investigated in a randomized, open-label, multi-centre trial, using PE as an active control (i.e. the feeder study: 16-HMedIdeS-12). A total of 30 subjects will be included in this study (20 in the imlifidase arm and 10 in the plasma exchange arm). The primary objective is to investigate the efficacy of imlifidase in removing DSA in patients who are experiencing an AMR episode after kidney transplantation.

While a rapid removal of DSA by imlifidase might be expected, DSA is likely to rebound unless well-controlled by concomitant immunosuppressive therapy. Therefore, there is also a need to address the long-term outcome of imlifidase as an AMR therapy. This will be studied during an extended follow-up period of 3 years in this study. Data for parameters such as kidney graft survival, patient survival, kidney function, treatment of rebound of donor specific antibodies (DSA) and anti-drug antibodies (ADAs) will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent obtained before any trial-related procedures
* Willingness and ability to comply with the protocol
* Previous treatment with imlifidase or plasma exchange in the trial 16-HMedIdeS-12

Note: The primary objective of this trial is overall graft survival after treatment with imlifidase or plasma exchange. Therefore, subjects can also be included even if the subject did not fully complete the feeder trial follow up but was dosed with imlifidase or plasma exchange in the trial 16-HMedIdeS-12.

Exclusion Criteria:

• Inability by the judgement of the investigator to participate in the trial for any other reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been treated with imlifidase or plasma exchange in the feeder study 16-HMedIdeS-12 may be included.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Operations, Study Director — Hansa Biopharma AB
Locations (7):
- Universitätsklinik für Innere Medizin III, Klinische Abteilung für Nephrologie MUW, Vienna, Austria
- France (4):
  - Hôpital Pellegrin, Bordeaux
  - CHU Grenoble Alpes - Néphrologie, dialyse et transplantation, Grenoble
  - Hôpital Saint-Louis. Service de Néphrologie et Transplantation, Paris
  - Hôpital Necker - Service de Néphrologie - Transplantation, Paris
- Germany (2):
  - Charité-Universitätsmedizin. Dept. of Nephrology and Medical Intensive Care, Berlin
  - Medizinische Hochschule Hannover, Hanover

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Halleck F, Bohmig GA, Couzi L, Rostaing L, Einecke G, Lefaucheur C, Legendre C, Montgomery R, Hughes P, Chandraker A, Wyburn K, Halloran P, Maldonado AQ, Sjoholm K, Runstrom A, Lefevre P, Tollemar J, Jordan S. A Randomized Trial Comparing Imlifidase to Plasmapheresis in Kidney Transplant Recipients With Antibody-Mediated Rejection. Clin Transplant. 2024 Jul;38(7):e15383. doi: 10.1111/ctr.15383. PMID 39023092

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12
Started | 11 | 7
Completed | 3 | 1
Not Completed | 8 | 6
Not completed — Graft loss | 2 | 1
Not completed — Patient not eligible as no AMR in feeder trial | 1 | 0
Not completed — Study terminated by sponsor | 5 | 3
Not completed — Sponsor decision | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12 | Total
Number analyzed (Participants) | 11 | 7 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.9 (17.6) | 48.0 (13.5) | 46.7 (15.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 4 | 9
  Male | 6 | 3 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 8 | 6 | 14
  Asian | 0 | 1 | 1
  Black or African American | 3 | 0 | 3
Region of Enrollment [Number; unit: participants]
  Austria | 1 | 3 | 4
  France | 8 | 2 | 10
  Germany | 2 | 2 | 4
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27.1 (6.9) | 29.0 (7.1) | 27.8 (6.8)

OUTCOME MEASURES:

1. Primary Outcome: Overall Graft Survival at Year 3
Description: Graft survival is defined as time from start of AMR treatment in feeder study (16-HMedIdeS-12) to graft loss. Graft loss is defined as permanent return to dialysis for at least 6 weeks, re-transplantation, or nephrectomy.
  Data table show number of patients with a functioning graft at Year 3.
Time Frame: 3 years after start of AMR treatment in feeder study (16-HMedIdeS-12)
Population: Due to the premature termination of the trial, 7 patients in the Imlifidase treatment group and 6 patients in the Plasma exchange treatment group had no graft survival data for the 3 year timepoint
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12
Number analyzed (Participants) | 11 | 7
Participants
  Number of patients with a functioning graft | 2 | 0
  Number of patients with graft loss | 2 | 1
  Censored (patients being censored up to the time point) | 7 | 6

2. Secondary Outcome: Overall Graft Survival at Year 2
Description: Graft survival is defined as time from start of AMR treatment in feeder study (16-HMedIdeS-12) to graft loss. Graft loss is defined as permanent return to dialysis for at least 6 weeks, re-transplantation, or nephrectomy.
Time Frame: 2 years after start of AMR treatment in feeder study (16-HMedIdeS-12)
Population: Due to the premature termination of the trial, 6 patients in the Imlifidase treatment group and 4 patients in the Plasma exchange treatment group have no graft survival data for Year 2.
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12
Number analyzed (Participants) | 11 | 7
Participants
  Number of patients with a functioning graft | 3 | 2
  Number of patients with graft loss | 2 | 1
  Censored (patients being censored up to the time point) | 6 | 4

3. Secondary Outcome: Overall Graft Survival at Year 1
Description: as for outcome 2
Time Frame: 1 year after start of AMR treatment in feeder study (16-HMedIdeS-12)
Population: Due to the premature termination of the trial, 1 patient in each treatment group have no data for Year 1.
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12
Number analyzed (Participants) | 11 | 7
Participants
  Number of patients with a functioning graft | 8 | 5
  Number of patients with graft loss | 2 | 1
  Censored (patients being censored up to the time point) | 1 | 1

4. Secondary Outcome: Patient Survival at Year 3
Description: Overall patient survival is defined as time from start of AMR treatment in feeder study (16-HMedIdeS-12) to death for any cause.
Time Frame: 3 years after start of AMR treatment in feeder study (16-HMedIdeS-12)
Population: Due to the premature termination of the trial, 9 patients in the Imlifidase treatment group and 7 patients in the Plasma exchange treatment group have no survival data for the 3 year timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12
Number analyzed (Participants) | 11 | 7
Participants
  At risk (patients being at risk for event at the time point) | 2 | 0
  Event (patients having events up to the time point) | 0 | 0
  Censored (patients being censored up to the time point) | 9 | 7

5. Secondary Outcome: Kidney Function as Evaluated by eGFR
Description: Estimated glomerular filtration rate (eGFR) was calculated as described by the Modification of Diet in Renal Disease Study (MDRD) equation. eGFR is a measure of kidney function. eGFR for a kidney with normal function is 90 mL/min/1.72m2. Kidney disease is characterised by a decreased eGFR value.
Time Frame: 1, 2 and 3 years after start of AMR treatment in feeder study (16-HMedIdeS-12)
Population: Due to the premature termination of the trial a large proportion of the patients did not complete the trial and no data were collected for Year 3 in the "Plasma exchange treatment in feeder Study 16-HMedIdeS-12" arm.
Measure: Mean (Standard Deviation); unit: mL/min/1.73 m^2
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12
Number analyzed (Participants) | 11 | 7
mL/min/1.73 m^2
  Year 1: number analyzed (Participants) | 8 | 4
  Year 1 | 30.1 (20.9) | 36.6 (12.3)
  Year 2: number analyzed (Participants) | 3 | 1
  Year 2 | 41.2 (6.4) | 39.7
  Year 3: number analyzed (Participants) | 1 | 0
  Year 3 | 30.5 |

6. Secondary Outcome: Kidney Function as Evaluated by S/P-creatinine
Description: S/P-creatinine is a measure of kidney function. Kidney disease is characterized by an increased S/P-creatinine level.
Time Frame: 1, 2 and 3 years after start of AMR treatment in feeder study (16-HMedIdeS-12)
Population: Due to premature termination of the trial by the Sponsor, only very few patients had assessments at Year 2 and Year 3 and no data were collected for Year 3 in the "Plasma exchange treatment in feeder Study 16-HMedIdeS-12" arm.
Measure: Mean (Full Range); unit: umol/L
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12
Number analyzed (Participants) | 11 | 7
umol/L
  Year 1: number analyzed (Participants) | 8 | 4
  Year 1 | 297 [81 to 795] | 187 [102 to 288]
  Year 2: number analyzed (Participants) | 3 | 1
  Year 2 | 130 [107 to 161] | 187
  Year 3: number analyzed (Participants) | 1 | 0
  Year 3 | 144 |

7. Secondary Outcome: Number of Participants With Presumed or Biopsy Proven AMR Episodes
Description: Information about rejection episodes will be collected, according to Banff 2017 or later classification. For-cause biopsies together with contemporaneous local DSA analyses, kidney function parameters (creatinine, albumin/creatinine ratio in urine) and treatments (e.g. plasma exchange and IVIg) will be collected to assess the rejection episodes.
Time Frame: 3 years after start of AMR treatment in feeder study (16-HMedIdeS-12)
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12
Number analyzed (Participants) | 11 | 7
Participants | 9 | 6

8. Secondary Outcome: Number of Participants With Presumed or Biopsy-proven Rejection Episodes (Other Than AMR Episodes)
Description: as for outcome 7
Time Frame: 3 years after start of AMR treatment in feeder study (16-HMedIdeS-12)
Measure: Count of Participants; unit: Participants
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12
Number analyzed (Participants) | 11 | 7
Participants | 3 | 4

9. Secondary Outcome: DSA Levels
Description: DSA levels will be measured using single antigen bead human leukocyte antigen (SAB-HLA) assay
Time Frame: 1, 2 and 3 years after start of AMR treatment in feeder study (16-HMedIdeS-12)
Population: Due to premature termination of the trial by the Sponsor, some patients have no DSA assessments done at Year 1, Year 2 and Year 3 and no data were collected for Year 3 in the "Plasma exchange treatment in feeder Study 16-HMedIdeS-12" arm.
Measure: Mean (Standard Deviation); unit: Mean Fluorescence Intensity
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12
Number analyzed (Participants) | 11 | 7
Mean Fluorescence Intensity
  Visit 2 - feeder trial pre-treatment: number analyzed (Participants) | 10 | 5
  Visit 2 - feeder trial pre-treatment | 10764 (7603) | 15794 (5897)
  1 year post dosing: number analyzed (Participants) | 8 | 2
  1 year post dosing | 5964 (5539) | 3672 (643)
  2 years post dosing: number analyzed (Participants) | 3 | 1
  2 years post dosing | 2156 (1025) | 12362
  3 years post dosing: number analyzed (Participants) | 1 | 0
  3 years post dosing | 974 |

10. Secondary Outcome: ADA Levels
Description: The immunogenicity of imlifidase will be assessed by measuring ADA levels.
Time Frame: 1,2 and 3 years after start of AMR treatment in feeder study (16-HMedIdeS-12)
Population: Only patients exposed to imlifidase were assessed for anti-imlifidase antibodies (ADA).
  Due to premature termination of the trial by the Sponsor, some imlifidase treated patients have no ADA assessments done at Year 1, Year 2 and Year 3
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12
Number analyzed (Participants) | 11 | 0
mg/L
  1 year post dosing: number analyzed (Participants) | 8 | 0
  1 year post dosing | 75 (405) |
  2 years post dosing: number analyzed (Participants) | 3 | 0
  2 years post dosing | 41 (1426) |
  3 years post dosing: number analyzed (Participants) | 1 | 0
  3 years post dosing | 15 |

ADVERSE EVENTS:
Time Frame: From inclusion in the study until end of study (Year 3).
Description: Only AEs related to trial procedure or related to IMP administered in feeder trial were to be collected.
Arm/Group | Imlifidase Treatment in Feeder Study 16-HMedIdeS-12 | Plasma Exchange (PE) Treatment in Feeder Study 16-HMedIdeS-12
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/7
Other Adverse Events (participants affected / at risk) | 0/11 | 0/7

LIMITATIONS AND CAVEATS:
Early termination leading to small number of subjects analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the study, one or more manuscripts for joint publication may be prepared in collaboration between the investigator(s) offered authorship and Hansa Biopharma.

Any confidential information relating to imlifidase or the study, including any data and results from the study will be the exclusive property of Hansa Biopharma AB. The investigators and any other persons involved in the trial will protect the confidentiality of the proprietary information belonging to Hansa Biopharma AB

DOCUMENTS (2):
  • Study Protocol (2021-11-22): https://cdn.clinicaltrials.gov/large-docs/50/NCT04711850/Prot_000.pdf
  • Statistical Analysis Plan (2023-05-12): https://cdn.clinicaltrials.gov/large-docs/50/NCT04711850/SAP_001.pdf